CLINICAL TRIAL: NCT00002160
Title: A Multicenter Phase II/III, Placebo-Controlled Study of SNX-111 Administered Intrathecally to Cancer and AIDS Patients With Chronic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurex (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 256A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-03

CONDITIONS: HIV Infections; Cancer; Pain
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Pain; Palliative Care; omega-conopeptide MVIIA; Calcium Channel Blockers
MeSH Terms: conditions — HIV Infections; Neoplasms; Pain; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — ziconotide

INTERVENTIONS:
Drug: Ziconotide

SUMMARY:
To determine the safety and efficacy of SNX-111 in controlling severe, chronic pain in cancer and AIDS patients.

DETAILED DESCRIPTION:
Patients are randomized to receive SNX-111 or placebo (AS PER AMENDMENT 1/22/98: with randomization weighted 2:1 in favor of SNX-111) via external pump and an intrathecal catheter (thin tube inserted into the spinal canal). (AS PER AMENDMENT 1/22/98: the dose is increased every 24 hours, in the absence of onset of analgesia or adverse events. After 2-5 days, patients who respond to their medication continue treatment at home for 5-8 days. Patients who do not respond will be switched to the other regimen (i.e., placebo to SNX-111, or SNX-111 to placebo). After 10 days, responding patients are unblinded and asked to enroll in the long-term, open-label extension protocol. Patients remain on a fixed dose at the therapeutic level found in the previous study. The dose may be increased or decreased at the discretion of the investigator. Patients may continue therapy on a long-term basis until the drug is approved.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Rescue analgesia.

Patients must have:

* Chronic pain related to AIDS or cancer.
* Unsatisfactory response to prior opioid therapy.
* Life expectancy > 3 months (or 1 month if an infusion pump is in place).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Signs of sepsis or inadequately treated infection.

Patients with the following prior conditions are excluded:

History of heart disease, heart failure, or asthma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Ctr for Pain Management and Rehabilitation, Huntsville, Alabama
  - Gulf Coast Clinical Services, Mobile, Alabama
  - Northport Hosp, Northport, Alabama
  - Holt Krock Clinic, Fort Smith, Arkansas
  - Alta Bates Hosp, Berkeley, California
  - Pain Diagnosis and Treatment, Glendora, California
  - Univ of CA - San Diego, San Diego, California
  - Good Samaritan Hosp Ctr, San Jose, California
  - Connecticut Pain Care, Danbury, Connecticut
  - VA Med Ctr / Oncology Section, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - H Lee Moffit Cancer Ctr and Research Institute, Tampa, Florida
  - Emory Univ Hosp, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Pain Control Ctr, Chicago, Illinois
  - Elkhardt Gen Hosp, Elkhardt, Indiana
  - Neurosurgical Associates, Terre Haute, Indiana
  - Univ of Iowa Hosp, Iowa City, Iowa
  - Univ of Kansas Med Ctr, Kansas City, Kansas
  - New Orleans Pharmaceutical Research, Kenner, Louisiana
  - Louisiana State Univ, Shreveport, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Minneapolis Veterans Administration, Minneapolis, Minnesota
  - Univ of Missouri Med Ctr, Columbia, Missouri
  - The Pain Institute, Kansas City, Missouri
  - Cooper Hospital Early Intervention Program, Camden, New Jersey
  - Clinical Solutions, Princeton, New Jersey
  - Pain Management, New York, New York
  - Long Island Pain Management, Port Jefferson Station, New York
  - Univ of Rochester, Rochester, New York
  - Bowman Gray School of Medicine / Wake Forest Univ, Winston-Salem, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lehigh Valley Hosp, Allentown, Pennsylvania
  - Pennsylvania State College of Medicine, Hershey, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Methodist Hosp, Memphis, Tennessee
  - Univ of Tennessee, Memphis, Tennessee
  - Texas Tech Univ Health Science Ctr, Lubbock, Texas
  - Univ of Texas Health Sciences Ctr, San Antonio, Texas
  - Fairfax Hosp, Falls Church, Virginia
  - Swedish Pain Management, Seattle, Washington
  - Northwest Neuroscience Institute, Seattle, Washington
  - Marschfield Clinic, Marshfield, Wisconsin